CLINICAL TRIAL: NCT05847790
Title: Remote Pregnancy Monitoring to Improve Access: The REACTIVE Trial
Brief Title: Remote Pregnancy Monitoring to Improve Access
Acronym: REACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Samuel Parry, MD, Professor of OBGYN, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 852291
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-05

CONDITIONS: Fetal Monitoring
Keywords: Fetal monitoring; antenatal testing
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Remote NST (Experimental)
  Interventions: Device: Invu monitoring belt
- In-clinic NST - Standard of Care (Active Comparator)
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Invu monitoring belt — INVU monitoring belt used for remote NSTs
  Arms: Remote NST
Other: Standard of care — In-clinic NSTs - standard of care
  Arms: In-clinic NST - Standard of Care

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of remote nonstress test (NST) compared to in-clinic NSTs in improving fetal testing completion rates. Participants will be randomized to either in-clinic NSTs or use of an FDA-approved remote monitoring belt for their pregnancy monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age between 30 weeks 0 days and 35 weeks 6 days
* Pregnant patients who have clinical indication for fetal surveillance with NSTs (based on UPHS Health System clinical guidelines for antenatal monitoring)
* Able to provide written consent
* English speaking

Exclusion Criteria:

* Multiple gestations
* Maternal pre-gravid BMI greater than 45kg/m2
* Presence of an implanted pacemaker or defibrillator
* Active abdominal skin infection
* A known amniotic fluid index (AFI) less than 5cm or greater than 25cm on the most recent ultrasound (if available) prior to randomization
* Delivery is planned within 2 weeks of potential randomization

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Overall Fetal Testing Completion Rate | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  percentage of recommended antenatal testing sessions that were successfully completed as defined as a clinically interpreted test was performed
Fetal Testing Completion Rate in Black versus non-Black subjects | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Comparison between Black and non-Black subjects' percentage of recommended antenatal testing sessions that were successfully completed as defined as a clinically interpreted test was performed.

SECONDARY OUTCOMES:
Fetal Monitoring outcomes: Number of visits to the antenatal testing unit | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Count of visits to the office for in-person monitoring
Fetal Monitoring outcomes: Frequency of provider recommended prolonged monitoring | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Count of number of times provider recommends prolonged monitoring (defined by greater than 40 minutes of time on the monitor).
Fetal Monitoring outcomes: Time on NST monitor | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Sum of the number of minutes the subject is on the NST monitor
Fetal Monitoring outcomes: Number of non-reactive NSTs | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Count of the number of visits
Fetal Monitoring outcomes: Number of biophysical profiles performed for non-reactive NST tests | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Count of the number of biophysical profiles performed for non-reactive NST visits
Fetal Monitoring outcomes: Overall number of visits to the obstetrical triage unit | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Count of the number of visits to the obstetrical triage unit
Fetal Monitoring outcomes: Overall number of visits to the obstetrical triage unit directly related to a fetal monitoring visit | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Count of the number of visit directly related to an outpatient fetal monitoring appointment or session
Fetal Monitoring outcomes: Frequency of recommendation for delivery based on findings on fetal monitoring result | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Count of the number of subjects in each arm who receive a recommendation for delivery based on the findings of the fetal monitoring results.
Fetal Monitoring outcomes: Number of times a NST is not completed within the prescribed window | from 32 weeks gestational age to delivery, average of 10 weeks after enrollment.
  Count of number of NSTs which occur outside of prescribed window, for example, if a weekly testing regimen is prescribed, an appointment 8 or more days following the last one would count as 1 missed calendar window.
Obstetrics outcomes: Gestational age at delivery | time of delivery
  gestational age at time of delivery
Obstetrics outcomes: Number of participants with Preterm delivery | time of delivery
  preterm delivery is defined as less than 37 weeks gestational age
Obstetrics outcomes: Mode of delivery | time of delivery
  categorized as vaginal or cesarean
Obstetrics outcomes: Number of participants with an Indication for labor induction | time of labor induction
  in subjects who have labor induction, indication for inducing labor
Obstetrics outcomes: Number of participants with an Indication for cesarean section | time of delivery
  in subjects who have a cesarean section delivery, indication for cesarean section
Obstetrics outcomes: Composite neonatal morbidity score | from delivery to 6 weeks post-delivery
  Composite score of neonatal morbidity comprised of one or more of the following: severe respiratory distress, neonatal resuscitation outside of the delivery room, and death. This score could range from 0 to 3 with a higher score meaning a worse outcome
Obstetrics outcomes: Neonatal cord blood pH | time of delivery
Obstetrics outcomes: Apgar scores | five and ten minutes after delivery
  Apgar score at five and ten minutes after delivery, the score ranges from 0 to 10 with a higher score meaning a better outcome.
Obstetrics outcomes: Number of participants with an Admission to the neonatal intensive care unit | from delivery to 6 weeks post-delivery
Obstetrics outcomes: Admission to the neonatal intensive care unit for greater than 48 hours | from delivery to 6 weeks post-delivery
Obstetrics outcomes: Maternal length of stay | from delivery to discharge, up to 6 weeks post-delivery
Obstetrics outcomes: Neonatal length of stay | from birth to discharge, up to 6 weeks after birth
Cost-effectiveness outcomes: Productivity loss survey | at three timepoints, at time of randomization, 3 weeks after randomization (plus or minus 1 week) and 5 weeks after randomization (plus or minus 1 week)
  This survey will collect in half days increments the productivity impacts of the pregnancy, NSTs and for seeking health care for those reasons
Cost-effectiveness outcomes: Costs | from 32 weeks to delivery, average of 10 weeks after enrollment.
  Costs will be estimated based on collection of data on all health care visits, including outpatient, ED, OB triage and hospital admissions
Implementation outcomes: Theory-informed Acceptability Questionnaire | at time of delivery
  8-item Likert scale with range of values from 8 to 40 with a high score being more acceptable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States